CLINICAL TRIAL: NCT00555854
Title: Can a Behavioural Modifying Intervention Increase the Self-care and the Effect of the Diabetes Treatment in Chronically Ill Patients With Diabetes
Brief Title: Self-care Behaviour Treatment in Patients With Diabetes - a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 028; n
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes
Keywords: Motivational interviewing,; Multidisciplinary; Life style changes; Prevention; Compliance; Self Care; Behaviour
MeSH Terms: conditions — Diabetes Mellitus; Patient Compliance; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: An individual motivational intervention program to promote and maintain self-care behaviour — 5 individual interviews in an one year period

SUMMARY:
Diabetes is a common condition associated with increased morbidity and mortality. Non-pharmacological intervention strategies focusing on factors to improve self-management skills are considered an important part of the treatment in individuals with diabetes. Because of the increasing incidence in diabetes with costs (both physical, psychological and financial) for both patients and society it is important to investigate interventions that successfully promote self-care behaviour in patient with diabetes. Further research is needed to develop interventions effective in maintaining long-term glycemic control.

The aim of this project is to study the long-term effect of a motivational intervention program with an individual approach based on cognitive-behavioural strategies in chronically ill patients with diabetes. The effect will be evaluated on both physiological and psychosocial parameters including patient's experienced self-care competence.

The study will also provide an overview of what kind of non-pharmacological interventions that have been applied in relation to the treatment of type 2 diabetes and assess the effect of the various non-pharmacological interventions in randomised controlled trials.

DETAILED DESCRIPTION:
Diabetes is a common condition associated with increased morbidity and mortality. Non-pharmacological intervention strategies focusing on factors to improve self-management skills are considered an important part of the treatment in individuals with diabetes. Because of the increasing incidence in diabetes with costs (both physical, psychological and financial) for both patients and society it is important to investigate interventions that successfully promote self-care behaviour in patient with diabetes. Further research is needed to develop interventions effective in maintaining long-term glycemic control.

The aim of this project is to study the long-term effect of a motivational intervention program with an individual approach based on cognitive-behavioural strategies in chronically ill patients with diabetes. The effect will be evaluated on both physiological and psychosocial parameters including patient's experienced self-care competence.

The study will also provide an overview of what kind of non-pharmacological interventions that have been applied in relation to the treatment of type 2 diabetes and assess the effect of the various non-pharmacological interventions in randomised controlled trials; and identify factors shaping outcomes in the areas reviewed.

The hypothesis is that a motivational intervention program based on cognitive-behavioural strategies increases patient's belief in their own capability to succeed in their diabetes care and will lead to increased self-care behaviour changes in relation to diabetes.

Materials and Methods:

A randomized controlled trial with 400 patients with diabetes is carried out at an endocrinology unit in a Danish University Hospital. The sample size was determined by a power calculation based on a standard deviation of 1.15 in the HbA1c-value and a 5% two-sided significance level. The power is set to 90 %. Assessments are made at baseline, follow-up 1 year and follow-up 2 year. Statistical analysis will be used to compare end points between the two groups.

Focus group interviews with 15 patients from the interventions group are conducted. In order to investigate the participants lived experience of diabetes they are asked to talk about their experience of their daily life with diabetes, self-care activities and diabetes treatment. Data will be analyzed using a phenomenological approach.

To asses the effect of non-pharmacological interventions from previous randomised controlled trials a meta-analytic review is carried out. 40 studies are included in the analysis that had met the following inclusions criteria: 1) randomized controlled trials; 2) published in an English or Nordic language; 3) participants were adults with type 2 diabetes; 4) tested the effect of self-care behaviour interventions; 5) reported measures and statistical data on the effect of the intervention on diabetic specific parameters; and 6) information about means and standard deviations available to calculate effect sizes. The following databases were searched: Medline, PubMed, Embase, CINAHL, PsycInfo including PsychLIT, Cochrane Library and SveMed+. The effect sizes in the included studies will be pooled by use of a random-effects model because we expect heterogeneity between studies.

The perspective of the project is to increase the knowledge about non-pharmacological diabetes treatment to increase quality of life and the effect of survival for diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and female age above 18 years
* Diagnosed with diabetes completed and participated in a diabetes school program

Exclusion Criteria:

* Severe illness
* Cognitive dysfunction
* Not able to speak or read Danish
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2005-12; Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | one year

SECONDARY OUTCOMES:
Lipids profile ,blood pressure, waist, BMI and medication Questionnaire: PAID PCD HCCQ TSRQ Health Care Behavioural a | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, Ph.D, Principal Investigator — Institute of Clinical Research, University of Southern Denmark
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Rosenbek Minet LK, Wagner L, Lonvig EM, Hjelmborg J, Henriksen JE. The effect of motivational interviewing on glycaemic control and perceived competence of diabetes self-management in patients with type 1 and type 2 diabetes mellitus after attending a group education programme: a randomised controlled trial. Diabetologia. 2011 Jul;54(7):1620-9. doi: 10.1007/s00125-011-2120-x. Epub 2011 Apr 1. PMID 21455729